CLINICAL TRIAL: NCT03968237
Title: Measures to Improve Outcomes After an Opioid Overdose
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nassima Ait-Daoud Tiouririne (Other)
Responsible Party: Sponsor-Investigator, Nassima Ait-Daoud Tiouririne, Associate Professor, Director of UVA Center for Leading Edge Addiction Research, University of Virginia
Organization: University of Virginia (Other)
Other Study IDs: 21455
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine; Naloxone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Buprenorphine/Naloxone — Controlled substances
  Other Names: Belbuca; Probuphine; Narcan

SUMMARY:
This is a pilot study that aims to develop good clinical practices to improve outcomes after an opioid overdose and transition of care from the Emergency Department (ED) into an Office Based Opioid Treatment (OBOT) clinic for patients with opioid overdose/Opioid Use Disorder (OUD). We intend to involve UVA Emergency Medicine and Medical Toxicology physicians with buprenorphine waiver or an interest in becoming waived at our institution to implement early initiation of buprenorphine protocol. We hope that this change in practice will result in better management of patients with OUD and opioid overdose, reduce relapse and improve engagement in addiction treatment.

Subjects who meet criteria will be consented in the ED and receive a buprenorphine/naloxone induction protocol, prior to discharge and referral to the OBOT clinic. Subjects who consent to take part in this study will be entered in a database to track their involvement in treatment (s) at UVA and or any opioid related UVA health visits including OPIOID OVERDOSE.

DETAILED DESCRIPTION:
Every patient who is seen in the ED for opioid overdose and has received naloxone either by emergency medical services (EMS) or in the ED will be eligible to participate in this study. When patient is alert, they will be asked if they would be interested in participating in the study and consented when appropriate. Patients will receive a buprenorphine/naloxone induction protocol, prior to discharge and referral to the OBOT clinic.

OBOT Follow-up The patient's follow-up care will take place at the OBOT clinic, supervised by an Addiction Medicine specialist (physician) with a buprenorphine-waiver and an license clinical social worker (LCSW). Scheduling of all OBOT visits during this study are in alignment with the OBOT standard of care, including frequency and duration of visits. A total of 10 visits will be scheduled over the course of 6 months.

Month 1:

Visit 1:

The first OBOT visit will last approximately 60 minutes and will entail the following:

A standard initial evaluation, urine drug screen, urine pregnancy test, method of contraception, administration of the Brief Addiction Monitor (BAM), HIV-Risk Taking Behavior Scale, discussion of treatment plan and goals, and buprenorphine/naloxone prescription from physician.

Visits 2 through 4:

Each visit will last between 16 minutes to 1 hour. During each visit, the following tasks will be accomplished:

The subject will be asked about their drug use, urine drug screen, urine pregnancy test, method of contraception, discussion of treatment progress and adherence to plan and goals, therapy, and buprenorphine/naloxone prescription from physician.

Month 2:

Visits 5 and 6:

Each visit will last between16 minutes to 1 hour. During each visit, the following tasks will be accomplished:

The subject will be asked about their drug use, urine drug screen, urine pregnancy test, method of contraception, discussion of treatment progress and adherence to plan and goals, therapy, administration of BAM and HIV-Risk Taking Scale once (either of Visit 5 or 6), HIV-Risk Taking Behavior Scale and buprenorphine/naloxone prescription from physician.

Months 3 to 6:

Visits 7 through 10:

Each visit will last between 16 minutes to 1 hour. During each visit, the following tasks will be accomplished:

The subject will be asked about their drug use, urine drug screen, urine pregnancy test, method of contraception, discussion of treatment progress and adherence to plan and goals, therapy, administration of BAM and HIV-Risk Taking Scale, and buprenorphine/naloxone prescription from physician.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Person can read, write, and speak in English.
* Presenting to the University of Virginia ED with opioid overdose and administration of naloxone either by EMS or in the ED.
* Experiencing some withdrawal symptoms (COWS score of 12 or higher) or experiencing 3 of the following symptoms: tremor/twitching, irritability, joint or bone aches, bad chills or sweating, goose bumps
* Express an interest in receiving a buprenorphine/naloxone induction with the goal to continue the same treatment outpatient

Exclusion Criteria:

* Non-opioid substance overdose or overdose that does not respond to naloxone
* Patients requiring admission secondary to medical or psychiatric complications
* Patients on prescribed methadone
* Women who are pregnant; This medication may precipitate opioid withdrawal in pregnant patients with opioid use disorder. Withdrawal can harm the placenta function, preterm labor, fetal convulsions (seizures), stunted fetal growth and fetal death during pregnancy.
* Mothers who are breastfeeding
* Persons under the age of 18
* Persons not able to attend follow-up clinic visits
* Persons not able to consent
* Known allergy or sensitivity to buprenorphine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Emergency Room Department
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Opiate Withdrawal Scale (COWS) | at screening
  The COWS is an 11 item scale designed to be administered by a clinican. This tool is used to rate common signs and symptoms of opiate withdrawal and monitor these symptoms over time. Reduction in adverse events will be evaluated by the documentation of COWS scores right after administration of Naloxone, then buprenorphine/naloxone.
Opioid Related Emergency Department (ED) Visits | up to 30 days
  Reduce risk of opioid re-overdose following ED buprenorphine/naloxone induction protocol. This will be measured by calculating the percentage of opioid related visits to any ED at 7 days post discharge, at 30 days post discharge, and hospital admissions at 30 days discharge.
Treatment Engagement | up to 6 months
  Improve addiction treatment engagement for patients receiving ED buprenorphine/naloxone induction following opioid overdose. This will be measured by the number of ED patients scheduled for follow-up at the office based opioid treatment (OBOT) clinic versus number of patients that attend the scheduled first appointment and number of patients that continue to follow-up at the OBOT clinic at 30 days and at 6 months.

SECONDARY OUTCOMES:
Demographic Data | at screening
  The investigator will collect the demographic data of the population served by this protocol.
Brief Addiction Monitor (BAM) | up to 6 months
  Report of substance use and social and health outcomes. It is a 17 item, multidimensional questionnaire which assess three substance use disorder related aspects (risk factors for substance use, protective factors that support sobriety, and drug and alcohol use).
Urine Drug Screen | up to 6 months
  Percentage of urine toxicology positive for illicit drug and opioid use.
HIV Risk-Taking Behavioral Scale HIV Risk-Taking Behavioral Scale | up to 6 months
  Social and Health Outcomes. It is an 11 item validated scale for drug use and sexual behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Nassima Ait-Daoud Tiouririne, M.D., Principal Investigator — University of Virginia
Locations (1):
- UVA Center for Leading Edge Addiction Research, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No